CLINICAL TRIAL: NCT05979116
Title: Effect of Abdominal Myofascial Release on Pain and Functional Outcomes of Neck in Females with Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Khalil Mohamed Khalil, assistant lecturer, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004050
Record Dates: First submitted 2023-07-29; First posted 2023-08-07 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Cesarean Section
Keywords: cesarean section; myofascial release
MeSH Terms: interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: a single group study as a study that consists of only a single group of subjects included in the study design, in which all subjects received a single intervention and the outcomes are assessed over time .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- study group (Experimental): this study group will receive abdominal myofascial release
  Interventions: Other: myofascial release

INTERVENTIONS:
Other: myofascial release — MFR in its simplest form targeted restoration of mobility of myofascial and fascial layers from within, and with the surrounding structure. MFR techniques utilized with the cases include different variations of application: 1. Muscle was stroked in a long

SUMMARY:
To investigate the effect of abdominal myofascial release on pain, ROM and functional abilities of neck in females with CS scar.

DETAILED DESCRIPTION:
irty females with neck pain will participate in this study. Subjects will receive treatment session of thirty minutes in length in order to minimize tissue irritation and avoid increased tension of the scar area, which would counter the goal of the session.

Treatment sessions will be provided biweekly for two weeks apart in order to allow physiological and biomechanical healing time between treatment sessions.

MFR techniques will be employed to release the caesarean scar and myofascia of the DFL of each subject.

The depth of the scar in this study takes us through all the layers from the skin to the uterus, following the surgical incision procedure.

MFR was the primary treatment applied to the accessible structure of the patients' DFL, through Myers's MFR techniques of DFL. MFR in its simplest form targeted restoration of mobility of myofascial and fascial layers from within, and with the surrounding structure.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients suffering from chronic neck pain since more than 3 months.
2. They underwent CS since at least 2 year before entry into study.
3. Not suffering from neck pain before CS
4. Their age will range from 20 to 35 years.
5. They will be primiparous
6. Body mass index (BMI) will range from 20-30 kg/m2.

Exclusion Criteria:

1. Pregnancy.
2. BMI over 30 kg/m2.
3. Less than six months after CS.
4. History of pathologies resulting in weakening of connective tissue (diabetes, neoplasms, rheumatic illnesses).
5. Any abdominal surgeries other than caesarean sections.
6. Any head or neck trauma.
7. Skin irritation/inﬂammation at the site of scar.
8. Any spinal deformity as kyphosis or scoliosis.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
pain level measurement | 2 weeks
  The pain level of each subject will be assessed before participation and after the end of the treatment by using numerical rating scale. this scale have numbers from 0 to 10 with 0 means no pain at all and 10 means sever intolerable pain
Scar mobility | 2 weeks
  Subjects will lay supine on a plinth with arms at their sides and legs straight. Marks were made on the CS scar at 2.5 cm intervals. This resulted in from 5 to 8 measurement points along the scar, The examiner will use the marks to measure tissue extensibility in millimeters (mm) in each of four directions: superior/left/inferior/right by using adheremeter
pressure pain threshold measurement | 2 weeks
  Pressure pain threshold ( PPT) is defined as the force at which the subject asked for pressure to stop due to pain.
  The pressure algometer is an instrument used to assess PPT for musculoskeletal pain. It was used to measure PPT of neck muscles before and after the treatment program for each female.
  This device includes a 1 cm2 probe with a system to convert the force applied through a 1 cm2 pressure application surface to Newtons (N/cm2) or kilograms of force (kg/cm2), that appear on the display
Neck ROM | 2 weeks
  Neck ROM will be measured in a standardized sitting position to remove errors and movement compensation. The subjects will be asked for sitting with their back straight. Subject's ankles, knees and hips were positioned at right angle and arms were folded across the chest to minimize thoracic movement, with tongue depressor can be held between teeth for reference.
Functional disability index | 2 weeks
  The NDI is adapted from Oswestry Low Back Pain Disability Questionnaire. It consists of 10 questions: pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. 5 Each item is scored from 0 (no disability) to 5 (total disability).

CONTACTS AND LOCATIONS:
Overall Officials: Amel youssef, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chamorro Comesana A, Suarez Vicente MD, Docampo Ferreira T, Perez-La Fuente Varela MD, Porto Quintans MM, Pilat A. Effect of myofascial induction therapy on post-c-section scars, more than one and a half years old. Pilot study. J Bodyw Mov Ther. 2017 Jan;21(1):197-204. doi: 10.1016/j.jbmt.2016.07.003. Epub 2016 Jul 18. PMID 28167179
- [Background] Declercq E, Cunningham DK, Johnson C, Sakala C. Mothers' reports of postpartum pain associated with vaginal and cesarean deliveries: results of a national survey. Birth. 2008 Mar;35(1):16-24. doi: 10.1111/j.1523-536X.2007.00207.x. PMID 18307483
- [Background] Fan C, Guidolin D, Ragazzo S, Fede C, Pirri C, Gaudreault N, Porzionato A, Macchi V, De Caro R, Stecco C. Effects of Cesarean Section and Vaginal Delivery on Abdominal Muscles and Fasciae. Medicina (Kaunas). 2020 May 27;56(6):260. doi: 10.3390/medicina56060260. PMID 32471194
- See also: Effect of myofascial induction therapy on post-c-section scars, more than one and a half years old. Pilot study — http://pubmed.ncbi.nlm.nih.gov/28167179/
- See also: Mothers' reports of postpartum pain associated with vaginal and cesarean deliveries: results of a national survey — https://pubmed.ncbi.nlm.nih.gov/18307483/